# Uncovering Osteoporosis Clinical Trials: Firsthand Patient Insights Into Clinical Trial Experiences

# Informed Consent Form (ICF) For <u>Power Clinical Trial's</u> Osteoporosis Observational Study

Date: June 30, 2023

#### About the Informed Consent Document

Should you find yourself presented with this document, it signifies that you are being considered as a potential participant in an observational clinical trial centered around individuals with osteoporosis. In this, we thoroughly discuss the study, encompassing its objectives, execution plan, as well as potential benefits and drawbacks. Prior to making a decision about participation, it is essential to carefully assess your options and seek the counsel of a trusted confidant. In case any uncertainties or queries arise regarding the information provided, do not hesitate to approach the researcher for clarifications.

# Objectives of This Clinical Trial

Osteoporosis is a medical condition characterized by weakened and fragile bones. It occurs when the body loses bone mass or fails to produce enough new bone, leading to a decrease in bone density and structural integrity. As a result, the bones become porous, brittle, and susceptible to fractures even from minor impacts or stress.

Clinical trials for osteoporosis are designed to assess the safety and effectiveness of novel osteoporosis treatments. These trials play a crucial role in establishing whether these new treatments outperform existing options and provide substantial evidence to support their adoption within the wider population.

The primary aim of this particular study is to investigate the experiences of individuals diagnosed with osteoporosis who participate in a distinct clinical trial involving a medical

intervention. The focus will be on closely monitoring the rates of trial completion and withdrawal among these participants.

#### What it Means to Join an Observational Clinical Trial

In your role as a participant in this medical trial, you will become an integral part of an observational study—an insightful type of clinical trial aimed at gathering valuable information by closely observing individuals, without implementing any changes to their existing care plans.

During this trial, researchers will solely observe your progress and meticulously measure the outcomes of your condition, refraining from any form of intervention. This type of trial serves as a vital tool in attaining a deeper comprehension of the natural course of a specific condition and its impact on individuals who receive a diagnosis. By actively participating in this observational study, you will play a significant role in advancing medical knowledge and contributing to the enhancement of care for individuals who share the same condition.

## Exploring Osteoporosis Clinical Trials: A Comparative Analysis

There exists a diverse range of research goals when it comes to osteoporosis research. While this particular clinical trial adopts an observational approach, where specific treatments or interventions will not be administered, it is essential to recognize that other clinical trials for osteoporosis adopt an interventional nature, necessitating participants to undergo specific treatment protocols.

To make a well-informed decision regarding your potential participation in a clinical trial, it is vital to engage in thorough research and compare different studies. Valuable information regarding <u>osteoporosis studies</u> can be accessed through clinicaltrials.gov or by exploring Power's website, which provides details on currently open <u>osteoporosis</u> <u>clinical trials</u>. By investing time and effort into comprehending the various types of clinical trials available, you can confidently make a discerning decision regarding your suitability for trial participation.

Participating Voluntarily in Surveys for Clinical Trials

Exploring your experiences as a participant in this observational clinical trial is an integral part of our research. To gather this valuable information, we kindly request your participation in completing questionnaires every two weeks, which should take approximately 20-30 minutes of your time. Additionally, we will conduct check-in calls on a quarterly basis as long as you continue to be part of the trial.

It's crucial to emphasize that your involvement in the survey component of this trial is entirely optional. You have the autonomy to choose whether to answer all or some of the questions, and you retain the right to withdraw from the trial at any time if you wish. We understand that participation in a clinical trial is a personal decision, and we are committed to providing support throughout the process. Your privacy and comfort are of utmost importance to us, and we will fully respect your decision-making journey during the course of the trial.

### Maintaining Anonymity in Survey Responses

Preserving the confidentiality of your information is our highest priority throughout this clinical trial. To ensure your anonymity, we kindly request that you refrain from providing any personal or identifying details when responding to the questionnaires. The research team will take meticulous measures to protect your privacy. However, it is important to note that there may be specific legal circumstances under which the researcher is obligated to disclose your data.

# Benefits of Participating in an Observational Clinical Trial

While immediate benefits may not be evident for individuals participating in this observational clinical trial, their contribution holds the potential for a lasting impact on the lives of others. The valuable data gathered from participants will be utilized to improve the enrollment process for future osteoporosis patients, ensuring easier access to medical research opportunities. By actively joining this clinical trial, individuals have the opportunity to make a meaningful difference for future patients and play a vital role in advancing medical research.

Minimizing Risks: A Safe Approach in Observational Clinical Trials

Clinical trials have played a pivotal role in advancing the medical field, but it is crucial to acknowledge the potential health risks participants may face, particularly when novel treatments are involved. However, it is important to note that in our observational clinical trial, participants are not exposed to any new interventions, thereby eliminating such risks. Instead, participants are carefully observed, and outcomes are measured, ensuring their safety throughout the trial.

The confidentiality of participant information is a significant concern in clinical trials, and our medical study prioritizes safeguarding participant privacy. All data collected from participants is strictly anonymous, and access to this information is restricted solely to the research team.

Furthermore, stringent security measures are in place to protect all records, including call logs, online transactions, forms, and surveys. These records are securely stored with encryption and password protection, ensuring the confidentiality and privacy of participant information. These robust measures guarantee that participant information remains confidential and well-protected from unauthorized access, prioritizing the safety and privacy of all involved in the trial.

Exploring the Importance of Diversity in Clinical Trials: Further Research

For those interested in delving deeper into the subject of representation in clinical trials, there is a wealth of online resources available. These resources offer valuable insights into the challenges and opportunities surrounding diversity in clinical trials, providing a comprehensive understanding of the topic:

Clark, Luther T., Laurence Watkins, Ileana L. Piña, Mary Elmer, Ola Akinboboye, Millicent Gorham, Brenda Jamerson et al. "Increasing diversity in clinical trials: overcoming critical barriers." *Current problems in cardiology* 44, no. 5 (2019): 148-172.

Knepper, Todd C., and Howard L. McLeod. "When will clinical trials finally reflect diversity?." (2018): 157-159.

By consulting these resources, individuals can gain valuable knowledge to inform their own involvement in clinical trials and contribute to the advancement of diversity and inclusivity in research.

#### Confirmation of Informed Consent

I hereby confirm that I have devoted adequate time to thoroughly review and comprehend the contents of the informed consent form. I have undertaken this task independently or with the assistance of a trusted individual who has provided me with a comprehensive understanding of its contents. All queries and concerns I had have been effectively addressed, ensuring my complete satisfaction.

I am fully aware that my participation in this study is entirely voluntary, and I retain the right to withdraw my consent at any point, without the obligation to provide a justification or face any financial consequences. I have been duly informed that I will receive a copy of this informed consent form for my personal records.

Having meticulously considered and evaluated all the information presented to me, I willingly consent to participate in this study, exercising my own free will.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| <br>Date |

Acknowledgment by Consent Facilitator

As the consent facilitator, I affirm that I have thoroughly reviewed the contents of this document with the participant, ensuring a comprehensive understanding of the purpose, methods, potential risks and benefits, and other essential aspects of the osteoporosis clinical trial.

I have created a conducive environment for the participant to ask questions and seek clarification, addressing any confusion or misunderstandings that may have arisen. It is crucial to emphasize that the participant's involvement in this trial is entirely voluntary,

| and they retain the freedom to withdraw their consent at any time, without incurring any financial obligations. |
|---|
| Upon their expression of consent, I provided the participant with a copy of this document for their personal records. |
| Printed Name of Person Taking Consent |
| Signature of Person Taking Consent |
| Date |